CLINICAL TRIAL: NCT01770067
Title: Prospective Evaluation of the Efficacy and Safety of Continuous In-situ Ultra High-dose Antibiotics (CITA) and Minimally Invasive Surgery (MIS) Utilizing Regulated Negative Pressure-assisted Wound Therapy (RNPT) in the Salvage of Infected Cardiovascular Implantable Electronic Devices (CIED) by Localized High-dose Antibiotics
Brief Title: Salvage of Infected Cardiovascular Implantable Electronic Devices (CIED) by Localized High-dose Antibiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0093-12-HYMC
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Infection
Keywords: Cardiac Resynchronization Therapy Devices
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infected CIED and Infection-Prone Patients Prior to CIED Implantation (Experimental): Administration of high-dose antibiotics (CITA)
  Interventions: Drug: CITA-RNPT
- Infected CIED extraction (Active Comparator): Extraction of infected CIED
  Interventions: Procedure: Extraction of infected CIED

INTERVENTIONS:
Drug: CITA-RNPT
  Arms: Infected CIED and Infection-Prone Patients Prior to CIED Implantation
Procedure: Extraction of infected CIED
  Arms: Infected CIED extraction

SUMMARY:
Following previous positive experience with regulated CITA-RNPT of infected CIEDs, we suggest increasing the number of recruited patients and that CITA-RNPT can be administered prophylactically to patients prior to replacement of previously treated CIEDs, immuno-compromised patients, and others.

ELIGIBILITY:
Inclusion Criteria:

* High-risk patients for CIED infections
* CIED infections

Exclusion Criteria:

* Systematic infection

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Lack of CIED Infection | One year

CONTACTS AND LOCATIONS:
Overall Officials: Moris Topaz, MD, PhD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Topaz M, Chorin E, Schwartz AL, Hochstadt A, Shotan A, Ashkenazi I, Kazatsker M, Carmel NN, Topaz G, Oron Y, Margolis G, Nof E, Beinart R, Glikson M, Mazo A, Milman A, Dekel M, Banai S, Rosso R, Viskin S. Regional Antibiotic Delivery for Implanted Cardiovascular Electronic Device Infections. J Am Coll Cardiol. 2023 Jan 17;81(2):119-133. doi: 10.1016/j.jacc.2022.10.022. PMID 36631206